CLINICAL TRIAL: NCT01103154
Title: A Controlled Trial of Nadolol Plus Isosorbide Mononitrate vs. Carvedilol for the Prevention of Variceal Rebleeding
Brief Title: A Trial of Nadolol Plus Isosorbide Mononitrate Versus Carvedilol for the Prevention of Variceal Rebleeding
Acronym: Carvedilol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: E-DA Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Gin-Ho Lo, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Carvedilol vs. N+I; vghks96CT2-13 (Other: vghks96CT2-13)
Record Dates: First submitted 2010-04-09; First posted 2010-04-14 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Variceal Rebleeding
Keywords: beta blocker; variceal rebleeding; efficacy and safety in reducing variceal rebleeding
MeSH Terms: interventions — Carvedilol; Nadolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol (Active Comparator): carvedilol 6.25mg per day
  Interventions: Drug: carvedilol
- N+I (Active Comparator): nadolol 40mg per day, ISMN 10 mg per day
  Interventions: Drug: nadolol + ISMN

INTERVENTIONS:
Drug: carvedilol — 6.25mg per day, increase to 6.25mg bid
  Arms: Carvedilol
Drug: nadolol + ISMN — nadolol 40-80mg ISMN 10-20mg
  Arms: N+I

SUMMARY:
Carvedilol is shown to be superior to propranolol to reduce the portal pressure. This study was undertaken to compare the effectiveness and complication rates of nadolol and isosorbide mononitrate (ISMN) with carvedilol in the prevention of rebleeding from esophageal varices.

DETAILED DESCRIPTION:
Bleeding from esophageal varices is a severe complication of portal hypertension. After initial control of acute variceal bleeding, patients have up to a 70% risk of rebleeding. Of those do rebleed, there is a 20%-35% mortality rate. Therefore, preventive procedures are required for patients surviving an episode of acute variceal bleeding. Both endoscopic injection sclerotherapy (EIS) and propranolol have been well documented to be effective for the prevention of variceal rebleeding. In recent years, endoscopic variceal ligation (EVL) has replaced EIS as the endoscopic treatment of choice in the management of bleeding esophageal varices. On the other hand, the addition of isosorbide-5-mononitrate (ISMN) has been shown to be even more effective than propranolol alone in the reduction of portal pressure and in the prevention of variceal rebleeding. A controlled trial showed that the combination of nadolol and ISMN was better than EIS in terms of prevention of variceal rebleeding and complications. The combination of nadolol and ISMN has been shown to be better than EVL in preventing variceal rebleeding. However, our study showed a contradictory result. On the other hand, carvedilol is shown to be superior to propranolol to reduce the portal pressure. This study was undertaken to compare the effectiveness and complication rates of nadolol and ISMN with carvedilol in the prevention of rebleeding from esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

1. acute or recent bleeding from esophageal varices (defined below),
2. the etiology of portal hypertension was cirrhosis, and
3. age was between 20 and 70 years old.

Exclusion Criteria:

1. association with hepatocellular carcinoma or other malignancy,
2. association with cerebral vascular accident, uremia, sepsis or other debilitating disease,
3. had history of gastric variceal bleeding,
4. received beta-blocker within 1 month prior to entry,
5. history of contraindication to the use of beta-blockers, such as asthma, heart failure, atrioventricular block, bradycardia (pulse rate <55/min) or arterial hypotension (systolic blood pressure < 90 mmHg),
6. history of prior shunt operation, TIPS (transjugular intrahepatic portosystemic stent shunt),
7. deep jaundice (serum bilirubin > 10 mg/dl),
8. encephalopathy greater than stage II,
9. failure in control of index variceal bleeding, or
10. refused to participate in the trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01

PRIMARY OUTCOMES:
variceal rebleeding | 2 years
  hematemesis or melena,requiring blood transfusion of 2 units or more bleeding source was proven endoscopically to be from esophageal varices

SECONDARY OUTCOMES:
adverse events, mortality | 2 years
  hypotension, bradycardia, dizziness, impotence, shortness of breath survival

REFERENCES:
- See also: National Health Research Institute, Taiwan — http://erad.nhri.org.tw/start